CLINICAL TRIAL: NCT05310370
Title: Correlation Between Homologous Recombination Deficiency Status and Resistance to PARP Inhibitors in Chinese Epithelial Ovarian Cancer Patients
Brief Title: HRD and Resistance to PAPPi in EOC Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: EOC-HRD3
Record Dates: First submitted 2022-03-26; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Epithelial Ovarian Cancer; Homologous Recombination Deficiency; Homologous Recombination Repair Gene Mutation; Poly(ADP-ribose) Polymerase Inhibitor; Drug Resistance; Progression-free Survival; Overall Survival
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A multiple panel testing of germline and somatic genes, including BRCA1/2, and HRD score are provided for all participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Testing of homologous recombination deficiency — A multiple panel testing of germline and somatic genes, including BRCA1/2, and HRD score are provided for all participants.

SUMMARY:
The association between homologous recombination (HR) gene mutations and homologous recombination deficiency (HRD) status in Chinese epithelial ovarian cancer (EOC) patients has been investigated in previous studies (NCT04190667 and NCT04651920). This study is to investigate the correlation between HRD and the resistance to poly(ADP-ribose) polymerase inhibitors (PARPi) in a Chinese cohort confirmed of epithelial ovarian cancer. The mutated genes, HRD score model and their relationship with the prognosis is the primary endpoint in this study. All enrolled patients will accept PARPi as maintenance therapy after the complete or partial remission of targeted lesions. A multiple panel testing of germline and somatic genes, including BRCA1/2, and HRD score are provided for all participants.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Pathological confirmation of epithelial ovarian cancer
* With available tumor tissues
* Given consents to participate the study
* With detailed follow-up outcomes

Exclusion Criteria:

* Not meeting all of the inclusion criteria
* Declining to accept PARPi as maintenance therapy after the major treatment for cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese cohort confirmed of epithelial ovarian cancer after the complete or partial remission of disease
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-03-26 (Actual); Primary Completion 2024-03-26 (Estimated); Study Completion 2025-03-26 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | One year
  Progression-free survival after the start of PARPi

SECONDARY OUTCOMES:
Overall survival | One year
  Overall survival after the start of PARPi
Severe adverse events | One year
  Severe adverse events after the start of PARPi

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China